CLINICAL TRIAL: NCT03777735
Title: Multicentric Observational Study on the Use of a Human Bone Graft in Osteochondral Defects
Brief Title: Human Bone Graft for Fixation of Osteochondral Defects in the Knee Joint
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Surgebright Gmbh (Industry)
Responsible Party: Principal Investigator, Catharina Chiari, Univ. Prof. Dr. Catharina Chiari, MSc, Medical University of Vienna
Other Study IDs: OD1
Record Dates: First submitted 2018-12-05; First posted 2018-12-17 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Osteochondral Defect
Keywords: human bone graft screw; osteochondral defect; knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- human bone graft screw: The patients will receive human bone graft screws surgically.
  Interventions: Procedure: human bone graft screw

INTERVENTIONS:
Procedure: human bone graft screw — All patients undergo surgical treatment of osteochondral defects in the knee joint with human bone graft screws.

SUMMARY:
This observational study is to document the application of a human bone graft in the surgical repair of bone fragment detachment in the knee joint (osteochondral defect) and its subsequent healing process.

DETAILED DESCRIPTION:
For the treatment of bone fractures metal screws have been used for decades. Removal of material is the major disadvantage of conventional osteosynthesis and requires a second intervention, with all the complications and risks for each patient. In order to avoid this second surgery, it is possible to use human bone screw grafts instead of metal screws.

The bone graft helps to create a solid, bony connection. This connection leads to an extension, a bone remodeling, bone installation and optimal reparation process in the affected area.

The comparatively rare occurrence of suitable patients contributes to the fact that there has not been enough systematic research to objectively confirm the benefits of the product, which is why this observational study is being conducted.

In total, 20 patients will be enrolled in several centers in Austria. The low number of cases and the multicenter design is due to the rarity of suitable patients.

This observational study will use Shark Screw® grafts without exception at all participating centers. These grafts are manufactured by two tissue banks, the Austrian Tissue Bank surgebright and the German Institute for Cell and Tissue Replacement (DZIG) and were approved by the competent Austrian authority (AGES) in 2016.

All patients participating in this observational study, due to a medical indication, undergo surgical treatment of osteochondral defects using the bone screws mentioned above.

Postoperatively, the patients are observed over a period of 24 months. In total, there are five follow-up examinations during which clinical examinations, x-rays and a magnetic resonance tomography (MRI) is performed. In addition the KOS-ADL and IKDC Score are collected.

ELIGIBILITY:
Inclusion Criteria:

* Indication for the use of a human bone graft in the surgical treatment of osteochondral defects
* legal capability of adults, guardians and adolescents aged 14 to 17 years, age-appropriate perceptivity for children 8 to 13 years old
* Written consent to participation in the study after previous written and oral education (additional consent for participation of minors in the study after prior written and oral education by at least one parent)
* Age ≥ 8 years

Exclusion Criteria:

* Insufficient knowledge of the German language
* Alcohol and drug abuse
* Pregnant or breastfeeding woman
* Foreseeable compliance issues
* Neoplastic diseases, malignant bone tumors, rheumatoid arthritis
* Active osteomyelitis
* Ulcerations in the area of the skin of the surgical area
* Immunosuppressive drugs that can not be discontinued

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from all participating sites scheduled for an OD treatment with human bone graft screws get information about this observational study and have the possibility to participate.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
incidence of surgical revisions | 1 year
  Was a surgical revision done postoperatively? YES/NO
incidence of loosening of the screw | 1 year
  based on x-rays or MRI: Is a loosening of the screw visible? YES/NO
incidence of cracking of the screw | 1 year
  based on x-rays or MRI: Is a cracking of the screw visible? YES/NO
incidence of loosening of the osteochondral fragment | 1 year
  based on x-rays or MRI: Is a loosening of the osteochondral fragment visible? YES/NO
incidence of cracking of the osteochondral fragment | 1 year
  based on x-rays or MRI: Is a cracking of the osteochondral fragment visible? YES/NO
time to healing of the osteochondral fragment | 1 year
  based on x-rays or MRI: Has the osteochondral fragment healed into the surrounding area? YES/NO
incidence of postoperative pseudoarthrosis | 1 year
  based on x-rays or MRI: Is a postoperative pseudoarthrosis visible? YES/NO
evaluation postoperative pain (VAS) | 1 year
  The visual analogue scale (VAS) is a vertical line, 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extremes (0mm = no pain - 100mm = worst imaginable pain). A higher score indicates more pain.
duration of postoperative job-related incapacity | 1 year
  evaluation of duration

SECONDARY OUTCOMES:
patient satisfaction (VAS) | 1 year
  The visual analogue scale (VAS) is a vertical line, 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extremes (0mm = very satisfied - 100mm = not satisfied at all). A higher score indicates less satisfaction.
Knee Outcome Survey - Activities of Daily Living Scale (KOS-ADL) | 1 year
  The KOS ADL score includes 14 questions and is divided in 2 subscales, symptoms (6 items, max. score 30) and functional restrictions (8 items, max. score 40). The scores of the answers range from 0 to 5 points. 0 points mean no impairment of everyday activities, while 5 points represent the greatest possible impairment. All points are summed up. From this, the KOS-ADL score is calculated as the proportion of the total response points from the possible maximum score (70) in percent. KOS ADL Score [%] = ( symptoms pts. + functional restrictions pts.)*100/70. The percentage ranges from 0-100%. 0% means no impairment, while 100% represents the greatest possible impairment.
International Knee Documentation Committee Subjective Knee Form (IKDC Score) | 1 year
  The IKDC Score contains 19 questions (7 questions for symptomatology, 10 concerning function, 2 about sport activity). The lowest function level or the highest symptom level receives the score value 1. The highest function level or the lowest symptom level is given the number n according to the number n of possible answers. With the exception of question 10 "Functioning before knee injury", the remaining 18 response points are summed up. This gives the "raw sum". The lowest possible score is 18 and the maximum possible score is 87. The raw sum is converted into a scale of 0 to 100 using the following formula: ((raw score - lowest possible score)/score range)*100. 0 points mean the greatest possible impairment, while 100 points mean complete freedom from symptoms and functioning. The IKDC score can only be calculated if at least 16 of the 18 questions have been answered.

CONTACTS AND LOCATIONS:
Overall Officials: Catharina Chiari, MD, Principal Investigator — Medical University Vienna
Locations (5):
- Austria (5):
  - LKH-Univ.Klinikum Graz, Graz
  - Barmherzige Schwestern Hospital Ried, Ried im Innkreis
  - General Hospital Vienna, Vienna
  - Orthopedic Center Otto-Wagner-Spital, Vienna
  - Hospital Wels- Grieskirchen, Wels

IPD SHARING:
Plan to Share IPD: No